CLINICAL TRIAL: NCT03797573
Title: Effects of Multichannel Transcranial Direct Current Stimulation to Reduce Hypertonia in Patients With Prolonged Disorders of Consciousness: a Pilot Study.
Brief Title: Multichannel tDCS to Reduce Hypertonia in Patients With Prolonged DOC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Aurore Thibaut, Principal Investigator, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014/280B
Record Dates: First submitted 2019-01-03; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Vegetative State; Minimally Conscious State; Spasticity, Muscle; Disorder of Consciousness
Keywords: transcranial direct current stimulation; disorder of consciousness; muscle hypertonia; spasticity; vegetative state; minimally conscious state
MeSH Terms: conditions — Persistent Vegetative State; Muscle Spasticity; Consciousness Disorders; Muscle Hypertonia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS (Active Comparator): Patients will receive tDCS (bilateral fronto-central stimulation) during 20 minutes preceded and followed by a clinical assessment (Modified Ashworth Scale and Coma Recovery Scale-Revised) and neurophysiological assessment (8 channels EEG).
  Interventions: Device: tDCS
- sham tDCS (Sham Comparator): Patients will receive sham tDCS (5 seconds of stimulation) during 20 minutes preceded and followed by a clinical assessment (Modified Ashworth Scale and Coma Recovery Scale-Revised) and neurophysiological assessment (8 channels EEG).
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: tDCS — tDCS will be applied during 20 minutes with a current of 1 mA preceded and followed by a behavioral assessments (Modified Ashworth Scale and Coma Recovery Scale Revised) and an EEG. The anodes will be placed over F3 and F4 and the cathodes over C3 and C4.
  Arms: active tDCS
Device: sham tDCS — Indentical to the active tDCS, except that the stimulation is terminated after 5 seconds.
  Arms: sham tDCS

SUMMARY:
Previous studies showed that transcranial direct current stimulation (tDCS) transiently improves performance of motor function in stroke patients, as well as decrease muscle hypertonia. In severely brain injured patients with disorders of consciousness (DOC), a single stimulation over the left dorsolateral prefrontal cortex has shown to improve patients' sign of consciousness. Nevertheless, other brain areas could be stimulated in order to manage other symptoms occurring in this population of patients, such as muscle hypertonia. In this study, investigators will assess the effects of bilateral fronto-central tDCS on spasticity as measured with the Modified Ashworth Scale (MAS) and on the Coma Recovery Scale-Revised (CRS-R) scores in patients with DOC in a double-blind sham-controlled experimental design.

DETAILED DESCRIPTION:
Following severe brain damage and coma, some patients may remain in a vegetative state (VS) or minimally conscious state (MCS). At present, there are no evidence-based guidelines regarding the treatment of patients with disorders of consciousness (DOC). A previous study showed that a single stimulation (using transcranial direct current stimulation - tDCS) of the left prefrontal cortex induces an behavioral improvement in some patients in DOC. Nevertheless, patients with DOC suffer from other invalidating dysfunctions such as spasticity (muscle hypertonia). In sroke patients, the inhibition of the motor cortex through cathodes placed over the motor region showed to reduce spasticity.

In this study, investigators aim to assess the effect of single session of transcranial direct current stimulation (tDCS) over right and left fronto-central areas (using 2 anodes and 2 cathodes), on the level of hypertonia and the level of consciousness of patients with DOC, in a double blind randomized sham controlled study. The anodes will be placed over F3 and F4, and the cathodes over C3 and C4.

tDCS is a form of safe non-invasive cortical stimulation, modulating cortical excitability under the electrodes, via weak polarizing currents. It has been reported that anodal tDCS transiently improves motor functions in healthy subjects and patients with stroke or Parkinson's disease.

By reducing the activity of the motor cortex (cathodes) and increasing the activity of the prefrontal cortex (anodes) we expect to observe a better motor function in patients with DOC.

ELIGIBILITY:
Inclusion Criteria:

* post comatose patients
* patients in minimally conscious state
* patients with stable condition
* patients free of sedative drugs and Na+ or Ca++ blockers (e.g., carbamazepine) or NMDA receptor antagonist (e.g., dextromethorphan)

Exclusion Criteria:

* premorbid neurology antecedent
* patients in coma
* patients < 28 days after the acute brain injury
* patients with a metallic cerebral implant
* cranioplasty
* shunt

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2014-06-28 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Change in MAS scores | baseline and directly after tDCS (20 minutes)
  Modified Ashworth Scale (MAS) will by assessed before and after tDCS (active and sham). Comparison of treatment effect (MAS score after tDCS minus before) between active and sham tDCS. The MAS is a 5 points scale going from 0 (no spasticity) and 5 (extreme spasticity).

SECONDARY OUTCOMES:
Change in the CRS-R total score | Baseline and directly after the tDCS (20 minutes)]
  Coma Recovery Scale Revised (CRS-R) will be performed before and after tDCS (anodal and sham). Comparison of the treatment effect (CRS-R total score score after tDCS minus before) between real and sham tDCS. The CRS-R is 23 points scale with 6 sub-scales (lower scores refer to reflexes, while higher scores refer to more complex behaviors). The total score is the sum of the scores in the 6 sub-scales.
Change in brain oscillations | Baseline and directly after the tDCS (20 minutes)
  8 channels electroencephalography (EEG) will be record before and after tDCS to record potential cortical changes induce by the stimulation. EEG power will be compared in different bandwidths (delta, theta, alpha, beta).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thibaut A, Bruno MA, Ledoux D, Demertzi A, Laureys S. tDCS in patients with disorders of consciousness: sham-controlled randomized double-blind study. Neurology. 2014 Apr 1;82(13):1112-8. doi: 10.1212/WNL.0000000000000260. Epub 2014 Feb 26. PMID 24574549